CLINICAL TRIAL: NCT01782105
Title: Intervention en Changement Des Habitudes de Vie Par l'Activité Physique et un Support Nutritionnel Durant la Grossesse en Estrie
Brief Title: Intervention to Promote Changes of Healthy Lifestyle (Physical Activity and Nutrition) During Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Diabetes Québec (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Marie-France Hivert, MD, MSc, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I-CHANGE
Record Dates: First submitted 2012-06-18; First posted 2013-02-01 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Excessive Weight Gain During Pregnancy; Gestational Diabetes
Keywords: weight gain; healthy lifestyle; gestational diabetes; adipokins; glycemic regulation
MeSH Terms: conditions — Diabetes, Gestational; Weight Gain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): In addition to the usual monitoring of pregnancy, this group will receive information about the recommended weight gain during pregnancy and an evaluation about of their nutritional and physical activity habits.
  Interventions: Behavioral: Control group
- Intervention group (Experimental): This group will receive a regular monitoring by health professionals (nutritionist and kinesiologist) who will ensure nutritional changes and physical activity necessary to secure the adoption of a healthy lifestyle and could participate to a physical activity group session once a week until week 36 of gestation.
  The intervention include:
  A nutritional counseling every 2 weeks by a nutritionist until week 36 of gestation; a physical activity group session once a week lead by a kinesiologist until week 36 of gestation; 2 sessions of physical activity counseling (weeks 12 and 24).
  Interventions: Behavioral: Healthy lifestyle counseling

INTERVENTIONS:
Behavioral: Healthy lifestyle counseling — Nutritionnal and physical activity counseling and physical activity session group
  Other Names: Intervention group
  Arms: Intervention group
Behavioral: Control group — Evaluation of nutritional and physcial activity habits
  Arms: Control group

SUMMARY:
The purpose of this study are:

* Assess the impact of an intervention to the adoption of healthy lifestyles among pregnant women at high risk of gestational diabetes mellitus on:

  * weight gain in pregnancy
  * the levels of maternal and fetal adipokines and
  * glycemic control maternal and fetal.
* Determine whether the adoption of healthy lifestyles in pregnancy is associated with epigenetic changes that influence the levels of adipokines and glucose regulation during pregnancy and in newborns.

ELIGIBILITY:
Inclusion Criteria:

* be aged ≥ 18 years,
* have a pre-pregnancy BMI ≥ 25 kg/m2,
* be at risk of developing a gestational diabetes mellitus (a history of gestational diabetes mellitus or glucose 1 hour post-50g > 7.1 mmol/L.

Exclusion Criteria:

* Pre-pregnancy diabetes detected in the first trimester (A1c > 6.5%, fasting glucose > 7.0 mmol/L, random blood glucose> 11.1 mmol/L, glucose > 10.3 mmol/L 1 hour post-50g)
* twin pregnancy
* taking medications that can affect blood sugar or weight,
* practice ≥ 150 minutes of physical activity per week
* against formal-indication for physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Weight change during pregnancy | Weeks 12, 24, 36 of gestation

SECONDARY OUTCOMES:
Levels of maternal and fetal adipokines | Weeks 12, 24 of gestation and at delivery (in cord blood)
Maternal and fetal glycemic control | Weeks 12, 24 of gestation and at delivery
  Results of glucose tolerance test (50g and 75g)
Determine whether the adoption of healthy lifestyle in pregnancy is associated with epigenetic changes that influence the levels of adipokines and glucose regulation during pregnancy and in newborns. | Weeks 12, 24 of gestation and at delivery (cord blood)
Optimize the intervention before measuring its impact on the prevention of gestational diabetes mellitus on a larger scale. | throughout the study
  Documentation will be collected about appreciation of the participants and attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Hivert, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada